CLINICAL TRIAL: NCT04031469
Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in Disease
Status: Suspended | Type: Observational
Why Stopped: Administrative
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-002
Record Dates: First submitted 2019-07-16; First posted 2019-07-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Gut Microbiome; Gastrointestinal Microbiome; Autism; Autism Spectrum Disorder; Autism Spectrum Disorder High-Functioning; Alzheimer Disease; Alzheimer Dementia (AD); Alzheimer Dementia; Alzheimer Disease (AD); Crohn; Crohn Colitis; Crohn Disease (CD); Crohn Disease Colon; Myalgic Encephalomyelitis; ME/CFS; Myalgic Encephalomyelitis (ME); Myalgic Encephalomyelitis/Chronic Fatigue Syndrome; Psoriasis; Psoriasis Annularis; Psoriasis Chronic; Chronic Urinary Tract Infection; Ulcerative Colitis (Disorder); Ulcerative Colitis (UC); Ulcerative Colitis Acute; Ulcerative Colitis Chronic; Multiple Sclerosis; Multiple Sclerosis (MS) - Relapsing-remitting; Multiple Sclerosis (MS) Primary Progressive; Constipation Chronic Idiopathic; Constipation; Celiac; Celiac Disease; Celiac Sprue; Lyme Arthritis; Lyme Borreliosis, Nervous System; Lyme Disease, Chronic; Cholesterol; Cholesterol Level, High; Cancer; Colon Cancer; Amyotrophic Lateral Sclerosis (ALS); Amyotrophic Lateral Sclerosis; Rheumatoid Arthritis (RA); Rheumatoid Arthritis - Rheumatism; Chronic Fatigue Syndrome (CFS); PARKINSON DISEASE (Disorder); Parkinson Disease; Parkinson Disease (PD); Depression; Major Depressive Disorder (MDD); Depression Disorder; Depression in Adults; Anxiety; Anxiety Disorder Generalized; Obsessive Compulsive Disorder (OCD); Obsessive Compulsive Disorder OCD; Obsessive - Compulsive Disorder; Bipolar; Bipolar 1 Disorder; Bipolar Disorder (BD); Bipolar Disorder I and II; Bipolar and Related Disorders; Migraine; Migraine Disorder; Diabetes (DM); Diabetes; Lupus; Lupus Erythematosus; Epidermolysis Bullosa (EB); Mesothelioma; Mesothelioma Malignant; IBS (Irritable Bowel Syndrome); Irritable Bowel; IBS - Irritable Bowel Syndrome; Irritable Bowel Syndrome (IBS); Eczema; Eczema Atopic Dermatitis; Acne; Myasthaenia Gravis; Gout
Keywords: Microbiome; autism; ASD; Myalgic encephalomyelitis; ME/CFS; Psoriasis; Chronic UTI; Chronic Urinary Tract Infection; Ulcerative Colitis; UC; Multiple Sclerosis; MS; Chronic Constipation; Constipation; Celiac disease; Celic Sprue; Lyme disease; Elevated Cholesterol; Colorectal Cancer; Cancer; Amyotrophic Lateral Sclerosis; ALS; Rheumatoid Arthritis; RA; Chronic Fatigue; Alzheimer disease; Chrohns colitis; Crohn; Alzheimer; Parkinson; depression; major depressive disorder; OCD; Obsessive-Compulsive disorder; Biopolar; Bipolar disorder; Migraine; Migraine headache; Diabetes; DM; Diabetes DM; Lupus; Lupus eruthematosus; Epidermolysis Bullosa; Mesothelioma; IBS; Irritable Bowel Syndrome; Eczema; Acne; Myasthenia Gravis; Gout
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Alzheimer Disease; Crohn Disease; Fatigue Syndrome, Chronic; Psoriasis; Colitis, Ulcerative; Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Constipation; Celiac Disease; Lyme Disease; Lyme Neuroborreliosis; Post-Lyme Disease Syndrome; Hypercholesterolemia; Neoplasms; Colonic Neoplasms; Amyotrophic Lateral Sclerosis; Arthritis, Rheumatoid; Parkinson Disease; Depression; Depressive Disorder, Major; Anxiety Disorders; Generalized Anxiety Disorder; Obsessive-Compulsive Disorder; Compulsive Personality Disorder; Bipolar Disorder; Bipolar and Related Disorders; Migraine Disorders; Diabetes Mellitus; Epidermolysis Bullosa; Mesothelioma; Irritable Bowel Syndrome; Eczema; Acne Vulgaris; Gout; Colorectal Neoplasms; Myasthenia Gravis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Stool samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- General Population: The general population will have their microbiome sequenced from stool samples provided.
  Interventions: Other: There is no intervention in this study

INTERVENTIONS:
Other: There is no intervention in this study — There is no intervention in this study

SUMMARY:
This study seeks to correlate microbiome sequencing data with information provided by patients and their medical records.

DETAILED DESCRIPTION:
The goal of this Research Study is to better understand how the genetic information in subject's microbiome correlates to the information provided in surveys and in medical records.

ELIGIBILITY:
Inclusion Criteria:

* 1. Signed informed consent, demonstrating that the patient understands the procedures required for the study and the purpose of the study
* 2. Male or female patients of any age (interest is given to children to compare with mothers).

Exclusion Criteria:

* 1. Refusal to sign informed consent form
* 2. History of bariatric surgery, total colectomy with ileorectal anastomosis or proctocolectomy.
* 3. Postoperative stoma, ostomy, or ileoanal pouch
* 4. Participation in any experimental drug protocol within the past 12 weeks
* 5. Treatment with total parenteral nutrition
* 6. Any clinically significant evidence of disease that could interfere with the subject's ability to enter the trial
* 7. Inability to adequately communicate with the investigator or their respective designee and/or comply with the requirements of the entire study

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and minors of any age
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2030-07-10 (Estimated); Study Completion 2030-12-10 (Estimated)

PRIMARY OUTCOMES:
Correlation of Microbiome to Disease via Relative Abundance Found in Microbiome Sequencing | One year
  Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the gut microbiome. These data will then be categorized among specific gastrointestinal disease types.

SECONDARY OUTCOMES:
Validation of Sequencing Methods | One year
  To validate the methods used to sequence samples

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Study Director — ProgenaBiome
Locations (1):
- Sabine Hazan, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hazan S, Stollman N, Bozkurt HS, Dave S, Papoutsis AJ, Daniels J, Barrows BD, Quigley EM, Borody TJ. Lost microbes of COVID-19: Bifidobacterium, Faecalibacterium depletion and decreased microbiome diversity associated with SARS-CoV-2 infection severity. BMJ Open Gastroenterol. 2022 Apr;9(1):e000871. doi: 10.1136/bmjgast-2022-000871. PMID 35483736